CLINICAL TRIAL: NCT03543475
Title: Cervical Pessary for Prevention of Spontaneous Preterm Birth in Singleton Pregnancies With Arrested Preterm Labor: a Randomized Controlled Trial
Brief Title: Cervical Pessary for Prevention of Spontaneous Preterm Birth in Singleton Pregnancies With Arrested Preterm Labor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: competing trial on same population.
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 103/18
Record Dates: First submitted 2018-04-30; First posted 2018-06-01 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pessary (Experimental): Silicon device applied on the cervix
  Interventions: Device: arabin pessary
- No Pessary (Active Comparator): standard care, no pessary
  Interventions: Device: no pessary

INTERVENTIONS:
Device: arabin pessary — arabin pessary: silicon device
  Arms: Pessary
Device: no pessary — control group
  Arms: No Pessary

SUMMARY:
Preterm birth (PTB) is a major cause of perinatal morbidity and mortality. Worldwide, about 15 million babies are born too soon every year, causing 1.1 million deaths, as well as short- and long-term disability in countless survivors.

Different strategies have been studied for prevention of spontaneous PTB (SPTB) in randomized controlled trials (RCTs), including progesterone, cerclage, cervical pessary, as well as lifestyle modification, such as smoking cessation, diet, aerobic exercise, and nutritional supplements. Most successful effort to reduce the incidence of SPTB have focused on asympatomatic women with risk factors, such as prior SPTB or short cervix. However, most SPTB occur in symptomatic women, i.e. women with preterm labor (PTL). Women with arrested PTL are at increased risk of SPTB.

The cervical pessary is a silicone device that has been used to prevent SPTB. The leading hypotheses for its mechanisms are two: that the pessary helps to keep the cervix closed, and that the pessary changes the inclination of the cervical canal so that the pregnancy weight is not directly above the internal os.

The aim of the study is to assess the efficacy of pessary in reducing preterm birth in women with arrested preterm labor

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestations
* Diagnosis of arrested PTL
* 18-50 years of age
* TVU CL ≤25mm at the time of randomization

Exclusion Criteria:

* Multiple gestations
* Rupture of membranes at the time of randomization
* Known major fetal structural (i.e. defined as those that are lethal or require prenatal or postnatal surgery) or chromosomal abnormality
* Fetal death at the time of randomization
* Cerclage in situ at the time of randomization
* Pessary in situ at the time of randomization
* Vaginal bleeding at the time of randomization
* Women who are unconscious, severly ill, mentally handicapped, or under the age of 18 years
* Placenta previa and/or accreta
* Ballooning of membranes outside the cervix into the vaginal or TVU CL = 0mm at the time of randomization
* Painful and regular uterine contractions at the time of randomization

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only pregnant women
Enrollment: 61 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Pre-term Birth | at the time of delivery
  delivery before 37 weeks of gestations

SECONDARY OUTCOMES:
Pre-term Birth <34, <32, and <28 weeks | at the time of delivery
  delivery before 34, 32, and 28 weeks
Mean gestational age at delivery in weeks | at the time of delivery
  Mean gestational age at delivery in weeks
Mean latency in days | at the time of delivery
  Time from randomization to delivery
Maternal side effects related to the intervention | at the time of delivery
  any maternal adverse events
Chorioamnionitis | at the time of delivery
  inflammation of the chorion and amnion by histopathological assessment after delivery
Composite adverse perinatal outcome | Between birth and 28 days of ag
  Includes Nectrotizing Enterocolitis, Intraventricular Hemorrhage, Respiratory Distress syndrome, Bronchopolmunary dysplasia,Retinopathy of Prematurity, Blood-culture proven sepsis, Neonatal death.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet

REFERENCES:
- [Derived] Mastantuoni E, Saccone G, Gragnano E, Di Spiezio Sardo A, Zullo F, Locci M; Italian Preterm Birth Prevention Working Group. Cervical pessary in singleton gestations with arrested preterm labor: a randomized clinical trial. Am J Obstet Gynecol MFM. 2021 Mar;3(2):100307. doi: 10.1016/j.ajogmf.2021.100307. Epub 2021 Jan 7. PMID 33422659